CLINICAL TRIAL: NCT03183492
Title: Long-term Persistence of Hepatitis A Immunity in Healthy Adults Vaccinated as Part of a Hepatitis A Universal Mass Vaccination Program
Brief Title: Immunogenicity and Persistence of GlaxoSmithKline (GSK) Biologicals' Havrix® in Healthy Adult Subjects Vaccinated at Infancy Under the Hepatitis A Universal Mass Vaccination (UMV) Program in Israel
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor cancelled the study as real life impact data has already shown the value of HepA vaccination & as no critical need to gather additional data in Israel.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 116762
Record Dates: First submitted 2017-05-30; First posted 2017-06-12 (Actual); Last update posted 2018-03-02 (Actual); Status verified 2018-03

CONDITIONS: Hepatitis A
Keywords: Israel; Universal Mass Vaccination; Havrix®; Hepatitis A; Healthy adults; Long term persistence; Toddlers
MeSH Terms: conditions — Hepatitis A | interventions — Hepatitis A Vaccines

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- HAV Group (Experimental): Subjects who were vaccinated under UMV with 2 doses of Havrix® Junior at infancy and will receive a single challenge dose of Havrix Adult at Visit 1 (Day 1).
  Interventions: Biological: Havrix®

INTERVENTIONS:
Biological: Havrix® — One challenge dose of Havrix® administered intramuscularly (IM) in the deltoid region of the non-dominant arm.
  Other Names: GSK Biologicals' inactivated hepatitis A vaccine

SUMMARY:
This study will evaluate the persistence, immunogenicity and safety of Havrix® (hepatitis A vaccine) in adults primed in infancy. The enrolled subjects will be assessed for circulating antibodies against hepatitis A and will also receive a challenge dose of Havrix Adult vaccine. In the present study, the anamnestic response will be assessed 30 days after the challenge dose.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who, in the opinion of the investigator, can and will comply with the requirements of the protocol
* Written informed consent obtained from the subject prior to performing any study specific procedure
* A male or female subject aged 18 to 19 years at the time of enrolment (up to but excluding the 20th birthday)
* Documented administration of 2 doses of Havrix® Junior in the second year of life
* Healthy subjects as established by medical history and clinical examination before entering into the study
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

has practiced adequate contraception for 30 days prior to study vaccine administration, and has a negative pregnancy test on the day of vaccine administration, and has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the study vaccine administration

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccine during the period starting 30 days before the dose of study vaccine (Day 29 to Day1), or planned use during the study period
* Any medical condition that in the judgment of the investigator would make intramuscular injection unsafe
* Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs during the period starting six months prior to the vaccine dose. For corticosteroids, this will mean prednisone ≥ 20 mg/day, or equivalent. Inhaled and topical steroids are allowed
* Administration of long-acting immune-modifying drugs at any time during the study entry
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product
* Administration of any hepatitis A vaccine dose, with the exception of the two doses of routine toddler vaccination for the subjects
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine
* Planned enrolment in the Israel Defense Forces within 30 days of study enrolment or activity that would prohibit the subject to return for Visit 2
* Acute disease and/or fever at the time of enrolment Fever is defined as temperature ≥38.0°C / 100.4°F. The preferred location for measuring temperature in this study will be the oral cavity Subjects with a minor illness without fever may be enrolled at the discretion of the investigator
* Pregnant or lactating female
* Female planning to become pregnant or planning to discontinue contraceptive precautions

Ages: 18 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2018-05-07 (Estimated); Primary Completion 2019-01-28 (Estimated); Study Completion 2019-01-28 (Estimated)

PRIMARY OUTCOMES:
Evaluation of immunity to hepatitis A in terms of anti-HAV (Antibodies against Hepatitis A virus) seropositivity status. | At the pre-challenge time-point (Day 1)
  A seropositive subject is a subject whose antibody concentration is greater than or equal to the cut-off value of 15mIU/mL.
Evaluation of immunity to hepatitis A in terms of anti-HAV antibody concentrations. | At the pre-challenge time-point (Day 1)
  Immunogenicity will be assessed in terms of Geometric Mean Concentration (GMC) of anti-HAV antibody concentrations.

SECONDARY OUTCOMES:
Evaluation of immunity to hepatitis A in terms of anti-HAV anamnestic response to hepatitis A vaccine challenge dose. | 30 days (Day 31) after challenge dose
  Anti-HAV anamnestic response to the challenge dose is defined as:
  At least a 4-fold increase in anti-HAV antibody concentrations in subjects seropositive at the pre-challenge time-point.
  Anti-HAV antibody concentrations at least 4 time the assay cut-off (i.e.60 mIU/mL) in subjects seronegative at the pre-challenge time-point.
Evaluation of immunity to hepatitis A in terms of anti-HAV seropositivity status in response to hepatitis A vaccine challenge dose. | 30 days (Day 31) after challenge dose
  A seropositive subject is a subject whose antibody concentration is greater than or equal to the cut-off value of 15mIU/mL .
Evaluation of immunity to hepatitis A in terms of anti-HAV antibody concentrations in response to hepatitis A vaccine challenge dose. | 30 days (Day 31) after challenge dose
  Immunogenicity will be assessed in terms of GMC of anti-HAV antibody concentrations.
Occurrence of solicited local and general symptoms. | During the 4-day (Days 1-4) follow-up period after the challenge dose
  The following local (injection-site) AEs will be solicited:
  Pain at injection site, Redness at injection site, Swelling at injection site.
  The following general AEs will be solicited:
  Fatigue, Fever*, Gastrointestinal symptoms**, Headache.
  *Fever is defined as temperature ≥38.0°C / 100.4°F. The preferred location for measuring temperature in this study will be the oral cavity.
  **Gastrointestinal symptoms include nausea, vomiting, diarrhea and/or abdominal pain.
  The AEs will be categorized depending on their intensity into the following grades:
  1. (mild) = An AE which is easily tolerated by the subject, causing minimal discomfort and not interfering with everyday activities.
  2. (moderate) = An AE which is sufficiently discomforting to interfere with normal everyday activities.
  3. (severe) = An AE which prevents normal, everyday activities.
Occurrence of unsolicited symptoms, according to the Medical Dictionary for Regulatory Activities (MedDRA) classification. | During the 31-day (Days 1-31) follow-up period after the challenge dose
  Unsolicited AE covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
Occurrence of Serious Adverse Events (SAEs). | After the challenge dose up to the study end (Days 1-31)
  SAEs to be assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of existing hospitalization, result in disability/incapacity or a congenital anomaly/birth defect in the offspring of a study subject.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.